CLINICAL TRIAL: NCT01564927
Title: Physiological Changes Associated With Deqi During Electroacupuncture to Right LI4 and LI11
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Yu Tai Wai David, Senior Physiotherapist, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSEARS20110510001
Record Dates: First submitted 2012-03-21; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: deqi electroacupuncture; BP HR HRV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electroacupuncture to right LI4 and LI11 (Experimental)
  Interventions: Device: Electroacupuncture to right LI4 and LI11 (ITO, EX-160)
- Electroacupuncture to knee caps (Sham Comparator): Electroacupuncture to knee caps
  Interventions: Device: Sham Electroacupuncture to knee caps
- Sham electroacupuncture to LI4 & LI11 (Placebo Comparator)
  Interventions: Device: Sham electroacupuncture to LI4 and LI11

INTERVENTIONS:
Device: Electroacupuncture to right LI4 and LI11 (ITO, EX-160) — Electroacupuncture at 2Hz, 0.4m/sec pulse duration
  Other Names: Electroacupuncture device, ITO, EX-160, Hannover, Germany
  Arms: Electroacupuncture to right LI4 and LI11
Device: Sham Electroacupuncture to knee caps — Electroacupuncture at 2Hz, 0.4m/sec pulse duration
  Arms: Electroacupuncture to knee caps
Device: Sham electroacupuncture to LI4 and LI11 — Electroacupuncture at 2Hz, 0.4m/sec pulse duration
  Arms: Sham electroacupuncture to LI4 & LI11

SUMMARY:
The aims of the study are to investigate the physiological responses associated with deqi during stimulation of the LI11 and LI4 acupuncture points and the correlation between the intensity of the deqi sensation to such responses.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy subjects who were naïve to acupuncture
2. Able to read Chinese and no communication barrier

Exclusion Criteria:

1. Subjects with medical disorders, including neurological and psychologic disorder
2. Use of medications that may affect the cardiovascular system within one week
3. Subjects with painful or uncomfortable sensations of upper and lower limbs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Physiological Changes Associated with Deqi during Electroacupuncture to Right LI4 and LI11 | One day
  heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: David TW YU, Master, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong, China